CLINICAL TRIAL: NCT00842439
Title: Biosocial Prediction and Intervention on Childhood Aggression
Brief Title: Healthy Brains & Behavior: Understanding and Treating Youth Aggression
Acronym: HBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 808689; SAP # 4100043366
Record Dates: First submitted 2009-02-02; First posted 2009-02-12 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Aggression
Keywords: aggression; Prevention and treatment of youth aggression
MeSH Terms: conditions — Aggression | interventions — Nuts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cognitive Behavioral Intervention (CBI) (Experimental): Participants will meet with an interventionist once a week for 12 weeks. They will discuss the child's behavior, will learn coping skills and how to deal with other people.
  Interventions: Behavioral: CBI
- Nutritional Supplements (NUT) (Experimental): Participants will be asked to take omega-3 supplements, multivitamin tablets, and calcium tablets every day for 12 weeks.
  Interventions: Dietary Supplement: NUT
- CBI + NUT (Experimental): Participants will receive both the cognitive behavioral intervention and the nutritional supplements.
  Interventions: Behavioral: CBI; Dietary Supplement: NUT
- No intervention (No Intervention): Participants will not be asked to come for sessions or any other intervention. They will receive a list of the types of help that are available if they are interested in following up on their own.

INTERVENTIONS:
Behavioral: CBI — Participants will have have one hour sessions, once a week for 12 weeks, where they will meet with an interventionist to go over cognitive-behavioral skills.
  Arms: CBI + NUT; Cognitive Behavioral Intervention (CBI)
Dietary Supplement: NUT — Participants will be asked to take omega-3 supplements, calcium tablets, and multivitamins every day for 12 weeks.
  Arms: CBI + NUT; Nutritional Supplements (NUT)

SUMMARY:
Understanding the joint neurobiological and social bases to aggression is critical to future attempts to tackle this major public health problem. The overarching goals are: (a) to conduct perhaps the most systematic integration of biosocial risk factors for childhood aggression in order to predict later aggression, (b) to conduct one of the very few biosocial interventions on childhood aggression, (c) to predict and treat two fundamentally different manifestations of aggression proactive and reactive aggression which likely have different etiologies and responsiveness to treatment. The specific aims are: (1) to assess biological (genetic, neurocognitive, brain imaging, neuroendocrinological, neurotoxin, psychophysiological, nutritional), psychosocial (neighborhood, family, school, peer, psychological) and psychiatric (ADHD, CD, ODD, depression, anxiety, PTSD, schizophrenia-spectrum) risk factors for male and female aggression in order to better predict later aggression, (2) to improve prediction by identifying the genetic, neuroimaging, psychophysiological, and neuroendocrinological factors that protect children who are socially at risk for a violence outcome, (3) to develop a genetic mouse model of aggression to test the effectiveness of nutritional interventions in reducing aggression, (4) to begin to develop a new biosocial approach to the treatment and prevention of aggression, based on both cognitive-behavioral and nutrition interventions, (5) to assess the differential prediction and treatment of two fundamental variants of child aggression: proactive and reactive aggression. The human sample will consist of 500 male and female 11-year-old children drawn from high-risk communities in Philadelphia. Three hundred participants will engage in a baseline assessment for risk factors for aggression, and then be randomly assigned to one of four three-month intervention programs: treatment-as-usual, cognitive-behavioral intervention, nutrition supplementation, or CBI + nutrition. Aggression outcome will be assessed throughout intervention and post-intervention.

The investigators believe that biological risk factors will interact with social risk factors in predicting aggression, over and above main effects of these classes of risk factors. Treatment effectiveness will interact with risk factors: those with low omega-3 and high lead exposure at intake will benefit most from the nutritional intervention; those with cognitive and affective risk factors will benefit most from the neuro-cognitive-behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

Entry into risk assessment component:

* Must be identified by their health care provider as meeting study criteria.
* Must be 11 or 12 years old
* Can be from the general population or who exhibit problem or aggressive behavior.
* Determination if the child meets criteria for enrollment into the at-risk risk group who will be entered into the RCT will be determined by the PI at the completion of the risk assessment day.
* Participant can be of any racial or ethnic background.
* Both youth and parent must be able to speak and understand English and able to provide informed assent/consent.

Entry into intervention component:

* Entry will be determined by the findings of the risk assessment that is conducted on study entry.
* Participants diagnosed with oppositional defiant disorder or have a borderline diagnosis
* Participants diagnosed with conduct disorder or have a borderline diagnosis
* Participants who score one standard deviation above the (normed population) mean on the either the reactive or proactive components of the Reactive-Proactive Aggression questionnaire
* Participants who score one standard deviation above the mean on the aggression subscale of the CBC, will be entered into the clinical trial
* These criteria may be relaxed slightly to ensure that we have sufficient participants in the intervention phase of the study.

Exclusion Criteria:

The goal is to be inclusive rather than exclusive, so as to achieve a more naturalistic cohort of community-residing children and their parent(s). Exclusion criteria are designed to deliberately limit the sample to eliminate, to the greatest possible extent, variables that might confound our primary aims.

Exclusion criteria include:

* A diagnosed psychotic disorder
* Mental retardation
* Claustrophobia
* Currently under psychiatric care
* Pervasive developmental disorders
* Conditions that preclude participation (or increase risk) in the clinical trial (Type 1 diabetes mellitus; metabolic diseases, gastro-intestinal disorders affecting nutrient absorption, cancer)
* Currently on medication that may modify lipid metabolism
* Extensive use of nutritional supplements within the previous 3 months
* Seafood allergy
* Presence or history of orthopedic circumstances and metallic inserts interfering with MR scanning; 11) pregnant in the case of females.
* There are no exclusions by sex or race/ethnicity.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 335 (Actual)
Dates: Start 2009-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic interviews and questionnaires will be used to see measure changes in aggression and antisocial behavior. We will also check for levels of Omega-3 before and after the interventions to see whether there are changes in Omega-3. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Raine, D.Phil., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Raine A, Gur RC, Gur RE, Richmond TS, Hibbeln J, Liu J. Omega-3 Supplementation Reduces Schizotypal Personality in Children: A Randomized Controlled Trial. Schizophr Bull. 2024 Aug 27;50(5):1117-1126. doi: 10.1093/schbul/sbae009. PMID 38300759
- [Derived] Raine A, Cheney RA, Ho R, Portnoy J, Liu J, Soyfer L, Hibbeln J, Richmond TS. Nutritional supplementation to reduce child aggression: a randomized, stratified, single-blind, factorial trial. J Child Psychol Psychiatry. 2016 Sep;57(9):1038-46. doi: 10.1111/jcpp.12565. Epub 2016 May 11. PMID 27166583